CLINICAL TRIAL: NCT03432351
Title: An International Multicenter Study of Isoelectric EEG Events in Infants and Young Children During Anesthesia for Surgery
Brief Title: Multi-center Isoelectric EEG Study in Children Under General Anesthesia
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Sydney Children's Hospitals Network (Other); Royal Children's Hospital (Other); Princess Margaret Hospital for Children (Other); Guangzhou Women and Children's Medical Center (Other); Yuying Children's Hospital of Wenzhou Medical University (Other); Sichuan Provincial People's Hospital (Other); Beijing Children's Hospital (Other); Shanghai Children's Medical Center (Other); Shengjing Hospital (Other); West China Hospital (Other); University of Geneva, Switzerland (Other); Erasmus Medical Center (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-014608
Record Dates: First submitted 2018-01-02; First posted 2018-02-14 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Electroencephalography; General Anesthesia; Pediatric Anesthesia
Keywords: EEG; Electroencephalography; Pediatric anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children: 0-36mo: EEG sensor will be placed on the subject's forehead to observe and record EEG activity. No other applicable intervention.

SUMMARY:
Multi-center, prospective, observational study investigating the incidence of isoelectric electroencephalography (EEG) events and the associated peri-operative factors in infants 0-3yo undergoing general anesthesia.

DETAILED DESCRIPTION:
Study will consist of placing a forehead EEG on the subject prior to induction of general anesthesia. EEG recording will continue until the end of anesthesia care. The anesthesiologist will be blinded to the EEG results during the study. Peri-operative factors such as demographics, vital signs, medications, etc... will also be recoded. Each site is expected to enroll up to 75 patients to provide at least 50 evaluable subjects. EEG files will be reviewed after recordings.

After informed consent has been obtained, the subject will receive standard anesthetic care as administered by the anesthesia provider, who will be blinded to the EEG display and data. EEG recording will continue until the end of anesthesia care.

After the recording, the EEG file will be reviewed and the number and duration of isoelectric events will be analyzed. Additional data that will be recorded include: patient demographic and perioperative factors (surgical procedure, anesthetic medications, end tidal anesthetic levels, induction and recovery room behavior, physiologic data, and time-stamps for intraoperative event. Post-operative questionnaire may also be sent to parents.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 to 36 (inclusive) months
* Greater than 36 weeks post-menstrual age (PMA) on the day of study
* Undergo general anesthesia for surgery that is expected to last more than 30 minutes (combined anesthesia and surgical time).
* Anesthetic maintenance with Sevoflurane if using volatile anesthetic or Propofol infusion if using total intravenous anesthetic.
* Expected airway management with a Laryngeal Mask Airway (LMA) or tracheal tube.
* Parental/legal guardian permission (informed consent) obtained

Exclusion Criteria:

* American Society of Anesthesiology (ASA) (physical status) greater than 3
* Structural/anatomical frontal brain malformations or other circumstances that make it difficult to apply the sensor to the forehead.
* History of abnormal EEG or severe neurological abnormalities.
* Scheduled for surgery above the neck, cardiac, brain, or emergency surgery.
* Known allergy or adverse reaction to ECG adhesives.
* On a sedative infusion (eg, propofol, morphine, fentanyl, midazolam, dexmedetomidine, ketamine) or recently on a sedative infusion (discontinued <24 hours ago)
* Received ketamine within 8 hours prior to the induction of general anesthesia

Max Age: 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 0-36 month old children undergoing general anesthesia for surgery.
Sampling Method: Probability Sample
Enrollment: 687 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Incidence of isoelectric EEG events in young children. | Up to 6 months after EEG recording
  Isoelectric EEG event is defined as low amplitude EEG for ≥ 2 seconds simultaneously across all 4 EEG channels.

SECONDARY OUTCOMES:
Discontinuity of isoelectric EEG events among age groups | Up to 12 months after EEG recording.
  Patient age associated with isoelectric EEG events will be analyzed using a Pearson Chi square test to compare discontinuity of isoelectric EEG events among the age groups
Association of isoelectric EEG events between gender groups | Up to 12 months after EEG recording
  Sample t-test or Wilcoxon rank-sum test, as appropriate will be used to analyze patient gender associated with isoelectric EEG events
Patient Weight associated with isoelectric EEG events | Up to 12 months after EEG recording
  Weight (kg)
Changes in patient's physical status associated with isoelectric EEG events | Up to 12 months after EEG recording
  Sample t-test or Wilcoxon rank-sum test, as appropriate, will be used to determine any association between the patient's physical status outcome associated with isoelectric EEG events.
Patient Gestational Age associated with isoelectric EEG events | Up to 12 months after EEG recording
  Gestational Age (weeks)
Procedure length associated with isoelectric EEG events | Up to 12 months after EEG recording.
  Procedure length (min)
Incidence of anesthetic type | Up to 12 months after EEG recording.
  Sample t-test or Wilcoxon rank-sum test, as appropriate, will be used to determine incidence of anesthetic type (gas vs. TIVA) associated with isoelectric EEG events.
Anesthesia dose | Up to 12 months after EEG recording.
  Sample t-test or Wilcoxon rank-sum test, as appropriate, will be used to determine variation in anesthesia dose associated with isoelectric EEG events.
Heart rate associated with isoelectric EEG events | Up to 12 months after EEG recording.
  Sample t-test or Wilcoxon rank-sum test, as appropriate, will be used to determine variation in heart rate (beats per minute) associated with isoelectric EEG events.
Blood pressure associated with isoelectric EEG events | Up to 12 months after EEG recording.
  Sample t-test or Wilcoxon rank-sum test, as appropriate, will be used to determine variation in blood pressure (mmHg) associated with isoelectric EEG events.
End tidal carbon dioxide (CO2) associated with isoelectric EEG events. | Up to 12 months after EEG recording.
  Sample t-test or Wilcoxon rank-sum test, as appropriate, will be used to determine variation in end tidal CO2 (mmHg) associated with isoelectric EEG events.
Anesthesia Recovery time associated with isoelectric EEG events. | Up to 12 months after EEG recording.
  Recovery time (min)
Changes in quality of life | Up to 2 months after EEG recording
  The patient's parent or guardian will complete the PedsQL questionnaire, which measures pediatric quality of life. It consist of up to 45 questions for a total score ranging from 0 to 180. The lower the total score, the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Hu, Study Director — Clinical Research Manager; Justin Skowno, Principal Investigator — Sydney Children's Hospitals Network; Andrew J Davidson, Principal Investigator — Royal Children's Hospital; Britta Regli-von Ungern-Sternberg, Principal Investigator — Princess Margaret Hospital for Children, Perth, Australia
Locations (15):
- United States (3):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
- Australia (3):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital (RCH, Melbourne, Australia), Parkville, Victoria
  - Princess Margaret Hospital for Children (PMH, Perth, Australia), Subiaco, Western Australia
- China (7):
  - Beijing Children's Hospital/Capital Medical University, Beijing, Beijing Municipality
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Jiao Tong university school of medicine / Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, China, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Erasmus MC Sophia Children's Hospital, Rotterdam, Netherlands
- University of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Coded limited dataset with minimum necessary protected health information (PHI) such as dates will be shared with Masimo and statisticians for EEG interpretation and data analysis.
Supporting Information: Study Protocol, SAP
Time Frame: Limited dataset will be available to other researchers for up to 2 years after end of study.